CLINICAL TRIAL: NCT06047704
Title: The Effect of State and Trait Anxiety on Pain-pressure Threshold
Status: Completed | Type: Observational
Sponsor: Philadelphia College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: H23024
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Pain; Anxiety; Musculoskeletal Pain; Sensitisation
MeSH Terms: conditions — Pain; Anxiety Disorders; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants-cross sectional: All participants received the same data collection protocol. No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The purpose of this research is to find out if different types of anxiety impact the sensation of how sensitive various muscles are to the application of pressure. This information can help researchers and healthcare providers better understand how people feel pain differently based on emotional factors This study is designed to study people who can be expected to have normal pain sensation processing

DETAILED DESCRIPTION:
Pain-Pressure threshold (PPT) measurements have been used extensively in both research and clinical practice. Its use allows for somewhat more quantifiable pain assessment and has been shown useful for discriminative validity in ruling in or out various conditions. (3) Individuals with higher scores on standardized measures of anxiety have been shown to be predisposed to lower (more sensitized) PPTs. As a part of medicines developing understanding of psychosocial variables in the experience of pain this relationship is consistent with other research findings.

Trait anxiety is an individual's tendency to appraise situations as threatening, avoid anxiety provoking situations, and demonstrate high baseline physiological arousal. State anxiety is defined as "transient state of arousal subjectively experienced as anxiety This research aims to measure the individual relationships that trait anxiety and state anxiety may have on PPTs. These findings may allow clinicians to better understand one element of the biopsychosocial model of pain.

Pain-Pressure threshold(PPT) testing is an increasingly common and accessible technique used by clinicians to gauge for potential altered sensory processing. While anxiety has been shown to impact PPT, research has not been published which aims to differentiate the roles of trait and state anxiety in modification of sensory processing. While trait anxiety is thought to be a longer-term characteristic, state anxiety is thought to be more transient and influenced by circumstances. Trait anxiety is thought to influence state anxiety but does not account for all presented state anxiety.

Research examining the potential impact of trait and state anxiety as distinct yet related constructs may allow providers to better extrapolate a patient's baseline pressure sensitivity with less unexplained variability based on potential state changes.

Subjects will begin with the completion of the STAI-5 with subscales for trait and state anxiety.

Next subjects will complete testing for pain-pressure thresholds at the bilateral upper trapezius and extensor carpi radialis muscles. Each site will be tested three times and the results averaged.

Pain pressure threshold testing will be performed in accordance with protocol parameters provided by the device manufacturer (Medoc) in conjunction with the pain-pressure threshold standardized protocol produced by the German Research Network on Neuropathic Pain (DFNS.) This device and protocol have been chosen due to high reliability and safety, with evidence to support their usefulness in research even for novice users. (6) Per the standardized instructions produced by the DFNS the subjects instructions will be as follows; "This is a test of your sensitivity to deep pressure. Now I will press this pressure gauge against your shoulder/forearm and will gradually increase the pressure. Please press the signal button provided to you as soon you would describe the pressure as 'slight discomfort.' Remember that this is not a pain tolerance test, it is a pain threshold test"

ELIGIBILITY:
Inclusion Criteria:

1) Adults 18 years of age or older 2: Able to read and complete the STAI-5 questionnaire as written in English

Exclusion Criteria:

1. pain lasting three months or longer, located anywhere in the body
2. severe health problems (such as cancer, cardiac, neurologic or psychiatric/anxiety disorders),
3. current pregnancy and/or gave birth in the last year.
4. Subjects currently taking medication which may impact sensory processing, such as antidepressants, opioids, neuroleptics, anticonvulsive drugs or steroids.
5. Subjects diagnosed with fibromyalgia or other conditions known to reduce muscular pain pressure thresholds, such as Lyme disease, polymyalgia, Lupus and Rheumatoid Arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers without exclusion reasons present
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Pain Pressure Threshold | Initial test with repeat measure at 21 days after
  Quantitative measurement of the amount of pressure applied at the point when the subject described the pressure as slight discomfort

SECONDARY OUTCOMES:
State-Trait Anxiety questionnaire (STAI)-Short form | Initial test with repeat measure at 21 days after
  A standardized test which measures both state and trait anxiety. Consists of two subscales, trait anxiety and state anxiety. Each section score ranges from 5 to 20, with a higher score indicating higher anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Philadelphia College of Osteopathic Medicine-GA, Suwanee, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
No IPD data sharing plan